CLINICAL TRIAL: NCT01799746
Title: Mechanisms of Response to Diesel Exhaust in Subjects With Asthma
Status: Withdrawn | Type: Observational
Why Stopped: The Airways Biology Initiative closed in December, 2015. This study was closed with the Penn IRB at that time. No subjects were recruited for this trial.
Sponsor: University of Pennsylvania (Other)
Collaborators: Rutgers University (Other)
Responsible Party: Sponsor
Other Study IDs: 817330
Record Dates: First submitted 2013-02-12; First posted 2013-02-27 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Other

SUMMARY:
In a controlled exposure setting, the study's goal is to determine the acute effect of diesel exhaust (DE) inhalation on airway inflammation and hyperresponsiveness (AHR) in subjects with mild to moderate stable asthma, using non-invasive measures.

DETAILED DESCRIPTION:
The investigators will also characterize selected polymorphisms in glutathione-S-transferase (GST) genes that have been implicated in susceptibility to air pollutants. Outcome measures will include lung function, bronchial responsiveness to bronchodilator, exhaled nitric oxide, induced sputum for inflammatory markers (IL6 and IL8), and exhaled breath condensate for nitrite, 8-isoprostane, 20-HETE (20-hydroxyeicosatetraenoic acid), nitrotyrosine and pH.

In this pilot project, parallel studies are being carried out in the human exposure chambers at two NIEHS centers, the EOHSI-CEED (Environmental and Occupational Health Sciences Institute- Center for Environmental Exposure and Disease) and the Penn-CEET (University of Pennsylvania-Center of Excellence in Environmental Toxicology). The joint project will enable each center to validate research results in a second population and include new biomarkers of pulmonary inflammation. Each center will recruit, consent, and collect data on its own subjects. Only de-identified data will be shared between the centers.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is an adult male or female between 18 and 55 years of age inclusive.
2. Subject must have a prior history of a physician's diagnosis of asthma with reversible airway obstruction (shown by a greater than 12% increase in FEV1 following bronchodilator; or a positive methacholine challenge done following the screening visit. If methacholine challenge is required for qualification, a physician will be on-site for the test. Subject's asthma has been stable for the past six months with no change in asthma therapy.
3. The subject has been a non-smoker for the past year and should have less than a 10-pack year history.
4. Subject must be free of other significant pulmonary diseases (i.e., cystic fibrosis, tuberculosis, interstitial lung disease and bronchopulmonary dysplasia.
5. The subject must be capable of and willing to provide written informed consent.
6. The subject is able to understand and comply with protocol requirements and timetables, instructions and protocol-stated restrictions.
7. The subject has no significant DE exposure that would include occupations such as truck driver, heavy equipment operator and railroad maintenance.

   -

Exclusion Criteria:

1. As a result of the medical interview, physical examination or screening investigations, the physician responsible considers the volunteer unfit for the study.
2. The subject has received an investigational drug or participated in any other research trial within 30 days or five half-lives or twice the duration of the biological effect of any drug (whichever is longer) prior to the current study.
3. Oral steroids within the last 6 months.
4. Less than 12% FEV1 response to bronchodilator or negative methacholine challenge.
5. Hospital admission for asthma in past 6 months.
6. The subject has a history of alcohol or drug abuse within the last 5 years.
7. The subject has history of hepatitis B, hepatitis C or HIV virus.
8. The subject has a history of cardiovascular disease including hypertension or says yes to one of the cardiovascular risk questions on the screening questionnaire.
9. The subject has a history of diabetes.
10. The subject is pregnant or lactating.
11. The subject has daily exposure to DE, i.e., trucking or heavy machine operators.

    -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All subjects will have been verified to meet criteria for mild/moderate asthma. At the same time all subjects will have been verified to be able to produce adequate sputum plugs for analysis.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
FEV1 response to bronchodilator, following DE compared with filtered air (primary outcome) | Up to 3 weeks

SECONDARY OUTCOMES:
Exhaled nitric oxide | Up to 3 weeks
8-isoprostane in exhaled breath condensate | 1 year
Nitrite in exhaled breath condensate | 1 year
pH in exhaled breath condensate | 1 year
20-HETE(20-hydroxyeicosatetraenoic acid)levels in exhaled breath condensate | 1 year
Cell differential in induced sputum | 1 year
Glutathione-S-transferase (GST)polymorphisms | Visit 1
Peak Flow | Up to 3 weeks
Forced Vital Capacity (FVC) | Up to 3 weeks
FEV1/FVC ratio | Up to 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Reynold A Panettieri, Jr., MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Airways Biology Initiative at Penn Presbyterian Medical Center, Philadephia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided